CLINICAL TRIAL: NCT03867591
Title: The Effect of Fermented Soy Supplementation on Occasional Heartburn Symptom Relief: A Randomized, Placebo-Controlled, Double-blind Trial
Brief Title: Fermented Soy and Heartburn Symptom Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Bio-Ingredients (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCR19814; IRB201900115 (Other: University of Florida)
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Heartburn; Acid Regurgitation
MeSH Terms: conditions — Heartburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study; the sponsor representative involved in the study, the investigator, the participants or site personnel involved in participant management or outcome assessment will remain blinded. Blinding to intervention will be used to reduce bias during data collection and evaluation of outcomes. At the investigational site, the randomization codes will remain secure at all times, but may be accessed in the event of an emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastro-AD® Group (Experimental): The participants randomized to this group 1 g of Gastro-AD® powder per sachet + flavoring agents.
  Interventions: Other: Gastro-AD®
- Placebo Group (Placebo Comparator): Participants in this arm will take a sachet containing maltodextrin (1 g) and exactly the same flavoring and coloring agents as Gastro-AD® powder flavored sachets.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Gastro-AD® — The product under study is Gastro-AD® fermented soy powder in the form of orodispersible flavored powder packed in non-transparent sachets.
  Content: 1 g of Gastro-AD® powder per sachet + flavoring agents.
  Arms: Gastro-AD® Group
Other: Placebo — The placebo product will have very similar appearance, color, texture and taste as the Gastro-AD® flavored sachet. The placebo sachets contain the respective amount of maltodextrin (1 g) and exactly the same flavoring and coloring agents as Gastro-AD® powder flavored sachets.
  Arms: Placebo Group

SUMMARY:
Heartburn is as common gastrointestinal symptom experienced by otherwise healthy adults and typically manifests as a painful burning sensation in the upper abdomen or in the chest. Typically, heartburn symptoms are treated with over-the-counter (OTC) medications which may come with side effects.

There is suggestive evidence of the efficacy of fermented soy (Gastro-AD®) for the heartburn symptom relief. The aim of the study is to evaluate the effect of a fermented soy on heartburn symptom relief and time to onset.

DETAILED DESCRIPTION:
Heartburn is as common gastrointestinal symptom experienced by otherwise healthy adults and typically manifests as a painful burning sensation in the upper abdomen or in the chest. Usually it is caused by the regurgitation of gastric acid into the esophagus. The prevalence of heartburn is 10-20% worldwide and is increasing. Typically, heartburn symptoms are treated with over-the-counter (OTC) medications which may come with side effects.

Gastro-AD® is a commercially available food supplement produced by fermentation of soy by a specific strain of Lactobacillus. There is suggestive evidence, in vivo as well as in vitro studies, of the efficacy of fermented soy (Gastro-AD®) for the heartburn symptom relief. The aim of the study is to evaluate the effect of a fermented soy on heartburn symptom relief and time to onset. It is hypothesized that the consumption of 1-3 g of fermented soy will relieve the heartburn symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent in English.
* Willing to have height and weight measured and provide demographic information (e.g. age, race, sex)
* Experience heartburn symptoms at least 2 days a week during the past 3 months.
* Use OTC product(s), supplements, or dietary manipulation to relieve heartburn symptoms in the last 3 months.
* Willing to take the study soy supplement before resorting to OTC product(s) to control heartburn symptoms.
* Willing to complete questionnaires, records, and diaries associated with the study and to complete all clinical visits.
* Willing to provide information about dietary intake; 3-day online 24-hr recalls during baseline, intervention, and washout.
* Willing and able to provide a valid social security for study payment purposes.

Exclusion Criteria:

* Do not meet the above criteria.
* Soy allergy
* Severe heartburn problem (cannot be ignored and often limits your concentration on daily activities) during the last week
* Diagnosed or currently being treated for any gastrointestinal diseases including GERD, gastric ulcers, Crohn's, celiac, ulcerative colitis, etc.
* Self-disclosed as pregnant or breast-feeding or planning on becoming pregnant during the study duration.
* Currently participating in another clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in severity of heartburn symptoms | 5 minutes, 15 minutes, 30 minutes
  Severity on a 5-point Likert scale ranging from 1 = no symptoms to 5 = severe discomfort

SECONDARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) | Baseline; Week 4; Week 5
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Change in Quality of Life (GERD-QOL) | Baseline; Week 4; Week 5
  The GERD-QOL is disease-specific instrument of 16 items combined into domains.
Heartburn event frequency | Baseline; Week 4; Week 5
  Heartburn events per period

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No